

Statistical analysis plan for the NEPNEP trial – a randomized controlled trial for chronic pain after primary total knee arthroplasty

Larsen, Jesper Bie; Skou, Søren Thorgaard; Laursen, Mogens; Bruun, Niels Henrik; Arendt-Nielsen, Lars; Madeleine, Pascal

<u>Publication date:</u>

17<sup>th</sup> January 2023

Document version:

1.0

# **Section 1: Administrative information**

## Title and trial registration

Item 1a: Descriptive title

Statistical analysis plan for the NEPNEP trial – a randomized controlled trial for chronic pain after primary total knee arthroplasty.

Item 1b: Trial registration number

Trial registration: ClinicalTrials.gov: NCT03886259 (registered 22.03.2019)

#### Version

Item 2: Statistical analysis plan (SAP version number with dates

Statistical analysis plan version 1.0. Date: 17<sup>th</sup> January 2023

#### **Protocol version**

Item 3:

The SAP is based on the protocol approved by the North Denmark Region Committee on Health Research Ethics (N-20180046) and the study protocol which was published the 24.02.2020 (1). The SAP was made publicly available prior to the last participant has completed the 12-month follow-up and before commencing any analyses of the outcomes.

## **SAP** revisions

Item 4a/b/c:

No revisions have been made

## Roles and responsibilities

Item 5: Roles, affiliations, and SAP contributors

Principal investigator:

Jesper Bie Larsen, PT, PhD, Musculoskeletal Health and Implementation, Department of Health Science and Technology, Faculty of Medicine, Aalborg University, Aalborg, Denmark

Study chair:

Søren Thorgaard Skou, PT, PhD, Professor, Research Unit for Musculoskeletal Function and Physiotherapy, Department of Sports Science and Clinical Biomechanics, University of Southern Denmark, Odense, Denmark, and The Research Unit PROgrez, Department of Physiotherapy and Occupational Therapy, Næstved-Slagelse-Ringsted Hospitals, Region Zealand, Denmark

Mogens Laursen, PhD, Orthopedic Surgery Research Unit, Aalborg University Hospital, Aalborg, Denmark

Niels Henrik Bruun, Unit of Clinical Biostatistics, Aalborg University Hospital, Aalborg, Denmark

Lars Arendt-Nielsen, PhD, Professor, Translational Pain Biomarkers, Department of Health Science and Technology, Faculty of Medicine, Aalborg University, Aalborg, Denmark

Pascal Madeleine, PhD, Professor, Sports Sciences – Performance and Technology, Department of Health Science and Technology, Faculty of Medicine, Aalborg University, Aalborg, Denmark

Item 6a: Signature of person writing the SAP

Date: 17.01.2023

ASKiv tekst her

Item 6b: Signature of senior statistician responsible

Jesper Bie Larsen

Item 6c: Signature of chief investigator

Jesper Bie Larsen

Date: 17.01.2023

### **Section 2: Introduction**

## **Background and rationale**

# Item 7:

Osteoarthritis is considered the most frequent cause of disability and pain in the elderly population, and the knee joint is one of the joints most commonly and severely affected(2,3). End-stage osteoarthritis is often treated with knee arthroplasty and primary total knee arthroplasty (TKA) is considered an effective treatment for pain relief and improved function(4,5). However, several studies have reported less favorable outcomes after primary TKA(6,7). Two systematic reviews found chronic pain rates after primary TKA of 13-17% among patients 12 months post-operatively and chronic pain rates at 2-7 years post-operatively varying between 8-27%(8,9). The causes of chronic pain after TKA remains largely unexplained(10). Signs of peripheral and central sensitization has been observed in chronic pain patients following TKA(10,11). The causes of chronic pain have been shown to be complex(12) and it has been suggested that the chronic pain in patients after TKA is predominantly centrally driven(10,11).

There is a lack of evidence-based treatments available for this group of patients. Therefore, this randomized controlled trial aims at investigating whether neuromuscular exercises combined with pain neuroscience education will provide superior results in terms of pain relief and improved physical performances compared to pain neuroscience education alone at 12-months follow-up.

## **Objectives**

Item 8: Description of objectives and hypothesis

The objective is to evaluate whether a 12-week neuromuscular exercise program combined with pain neuroscience education is superior to pain neuroscience education alone in terms of improving pain and physical performances at 12-months follow-up in a population of patients with chronic pain after primary TKA.

## Hypothesis:

We hypothesize that the patients randomized to neuromuscular exercise and pain neuroscience education will improve significantly more in pain and physical performances from baseline to 12-months than the patients randomized to pain neuroscience education alone.

### **Section 3: Trial methods**

### Trial design

Item 9: Description of trial design

This trial is designed as a randomized controlled superiority trial. Treatment allocation will be in a 1:1 ratio. The patients will be randomized to receive either neuromuscular exercises and pain neuroscience education or pain neuroscience education alone(1). The primary endpoint is at 12-months follow-up and a secondary endpoint, consisting of long-term follow-up, at 24-months.

#### Randomization

Item 10: Randomization details

The randomization was performed using computer-generated random numbers in permuted blocks of four to eight patients. After informed consent and baseline assessment had been conducted, the principal investigator randomly assigned patients to either of the treatment arms based on the computer-generated randomization. Thereafter, the allocation was provided to the patients.

The outcome assessors are blinded to the group allocation, are not a part of the provided interventions and are not affiliated with any of the treatment sites. Patients and physiotherapists providing the interventions cannot be blinded towards randomization.

### Sample size

Item 11: Full details of sample size calculation

For KOOS<sub>4</sub> and KOOS scores, a minimal clinically important difference of 10 is estimated, and commonly used(13). A sample size calculation was conducted to estimate how large a sample size is required to give the study a power of 90% to detect a minimum improvement of 10-point on the KOOS<sub>4</sub>, after 12 months follow-up, in the neuromuscular exercise and pain neuroscience education

group compared with the pain neuroscience education alone group (with a standard deviation of 15)(13,14). A two-sided significance level at 0.05 was set and results revealed that 49 patients are required in both groups. To account for possible missing data and a loss to follow-up of 20%, a total of 60 patients in each group was planned to be enrolled.

However, this study was impacted by the COVID-19 pandemic making recruitment particularly difficult and causing higher dropout rate than originally anticipated. Therefore, we were not able to recruit as many participants as planned and we decided to stop the trial early after recruiting for 44 months. Therefore, a total of 71 patients have been enrolled with 36 patients in the neuromuscular exercise and pain neuroscience education group and 35 patients in the pain neuroscience education alone group.

## Framework

Item 12: Description og hypothesis testing framework

All outcomes, i.e., primary, secondary, and other outcomes, will be evaluated in a superiority framework, hypothesizing that the patients receiving neuromuscular exercises and pain neuroscience education will improve more than patients receiving pain neuroscience education alone. A confidence interval including 10 points or more in the KOOS<sub>4</sub> score will be interpreted as a clinical meaningful difference, although we will interpret results with caution given the fact that we did not reach the target sample size.

# Statistical interim analysis and stopping guidance

Item 13:

No interim analysis was planned, and no adjustment of significance level was made. No stopping rules was defined a priory.

## Timing of final analysis

Item 14:

The analysis of primary, secondary, and other outcomes will be conducted collectively when all patients have reached the 12-month follow-up. The 12-month follow-up is expected to be finished in March 2023. An independent statistician (NHB) will conduct the analysis. Data from all time points (baseline, 3-, 6-, and 12-months) will be included in the analysis.

The analysis of the primary, pre-specified secondary and other outcomes (presented in item 26 and table 2) will be reported in the primary 12-month follow-up publication. Remaining secondary outcomes will be reported in subsequent, secondary publications.

Evaluation of long-term outcomes based on baseline to 24-months (including baseline, 3-, 6-, 12-, and 24-months) follow-up will be conducted when all patients have reached the secondary endpoint at 24-month follow-up and this data collection has ended.

### Timing of outcome assessments

Item 15:

All primary, secondary, and other outcomes will be evaluated at baseline, 3-, 6-, 12-, and 24-months, except for adverse events and adherence to interventions, which will be evaluated continuously during the intervention period and at 3-months, i.e., after the interventions have stopped. Further details can be found in the published study protocol(1)

## **Section 4: Statistical principles:**

# Confidence intervals and p-values

Item 16: Level of statistical significance

All conducted statistical tests will be two-sided and will be evaluated by a significance level of 5% (i.e., p=0.05).

Item 17: Description of planned adjustment for multiplicity

The NEPNEP trial has one clearly specified primary outcome and the secondary and other outcomes will serve as supportive and/or hypothesis generating, which is why multiplicity is not considered to be an issue (15).

Item 18: Confidence intervals

The presented confidence intervals will 95% and be two-sided.

### Adherence and protocol deviation

Item 19a: Definition of adherence to interventions

Adherence will be defined as participation in both pain neuroscience education sessions (valid for both groups). For the patients receiving neuromuscular exercises, adherence will be defined as participation in minimum 75% of the neuromuscular exercise sessions (i.e., 18 out of 24 exercise sessions). Adherence is registered by the physical therapists in charge of the neuromuscular exercise sessions and the pain neuroscience education sessions.

Item 19b: Description of how adherence to interventions will be presented

Adherence, for those randomized to neuromuscular exercise and pain neuroscience education, will be reported as the numbers and percentages of patients participating in at least 18 neuromuscular exercise sessions and participating in both pain neuroscience education sessions. Adherence, for those randomized to pain neuroscience education alone, will be reported as numbers and percentages of patients participating in both pain neuroscience education sessions.

Item 19c & 19d: Definition of protocol violation for the trial and how they will be presented

It is specified as an exclusion criterion if patients experience chronic pain due to loosening of implant or prosthesis failure which requires revision surgery. However, during the follow-up, patients might be referred to revision TKA surgery, e.g., based on new available information to the surgeon. Therefore, undergoing revision TKA during follow-up is defined as a major protocol

deviation, which could impact the outcomes of the trial. Number of patients in both randomized groups will be reported.

## **Analysis populations**

Item 20: Definition of analysis populations

All outcomes will be analyzed according to the intention-to-treat principles. The intention-to-treat population will be all subjects randomized to either group. A per-protocol analysis will be conducted based on patient adherence to interventions. Therefore, the following will be excluded from the per-protocol analysis: 1) The patients who did not participate in both pain neuroscience education sessions, 2) The patients in the neuromuscular exercises and pain neuroscience education group participating in below 75% (18 out of 24) of the neuromuscular exercise sessions and 3) patients receiving revision surgery at any time-point during follow-up.

# **Section 5: Trial population**

# Screening data

Item 21: Reporting of screening data

The recruitment period, from start date to end date, will be displayed as well as the total numbers of patients screened for eligibility throughout the recruitment period.

## **Eligibility**

Item 22: Summary of eligibility criteria

Patients were eligible to participate in the trial if they fulfilled the inclusion criteria:

- Male or female aged 40-80 years
- Body Mass Index (BMI) between 19-40 kg/m<sup>2</sup>
- Subjects with pain after primary TKA and  $\geq 12$  months post-operative
- For the index knee, duration of knee pain > 6 months.
- For the index knee, a perceived average daily pain score ≥ 4 (moderate-to-severe pain) over the last week prior to recruitment on a numerical rating scale (NRS, 0 (no pain) to 10 (maximum pain)).

Study exclusion criteria were:

- chronic pain due to loosening of implant or prosthesis failure requiring revision surgery
- secondary causes of arthritis to the knee, such as rheumatoid arthritis or sequelae from previous accidents
- surgery (including arthroscopy) of the index knee within three months prior to recruitment
- injury to the index knee within 12 months prior to visit
- acute pain, other than in the index knee, affecting the lower limb and/or trunk at the time of baseline testing
- participation in other pain trials two weeks prior to recruitment
- pregnancy
- drug and alcohol abuse

- rheumatoid arthritis, neurologic illnesses, or primary pain area other than knee (e.g., low back pain or upper extremity pain)
- lack of ability to adhere to protocol

#### Recruitment

Item 23 & 24: Information to be included in CONSORT flow diagram

A CONSORT flow diagram will be displayed, including the following information:

- Number of patients assessed for eligibility throughout the recruitment period
- Number of patients not meeting the inclusion criteria's or not consenting to participate
- Number of patients eligible for inclusion
- Number of patients randomized to both treatment arms
- Number of patients with follow-up assessment at 3-, 6-, 12-months for the primary analysis of 12-months follow-up<sup>1</sup>
- Number of patients with follow-up assessment at 3-, 6-, 12-, 24-months for the secondary long-term analysis of 24-months follow-up<sup>1</sup>
- Number of withdrawals or loss-to-follow-up for each timepoint and reasons for withdrawal or loss-to-follow-up
- Number of patients included in the intention-to-treat analysis and the per-protocol analysis

## **Baseline patient characteristics**

Item 25a: List of baseline characteristics to be summarized

Patients will be described with baseline, demographic characteristics which include age, sex, height, body mass, BMI, average daily pain intensity over last week, index knee, dominant leg, time-since-TKA-surgery, TKA in non-index knee, comorbidities, and scores on the Hospital Anxiety and Depression Scale(16). The following comorbidities will be recorded: Osteoarthritis in other areas than the index knee, chronic pain from other sites than the index knee, chronic obstructive pulmonary disease, diabetes, and cardiovascular disease. Comorbidities will be registered using the medical journals.

Item 25b: Details on how baseline characteristics will be descriptively summarized

Table 1 illustrates how the baseline characteristics will be presented. Continuous data will be presented as mean and SD if data is normal distributed and as median and range if data is non-normal distributed. Categorical data will be presented as numbers and percentages. No test for statistical significance for the baseline characteristics will be conducted in line with recommendations by the CONSORT statement (17). Instead, the clinical importance of any imbalances will be considered.

 $<sup>^{1}</sup>$  Number of patients with follow-up assessment is defined as patients with data available for the primary outcome (KOOS<sub>4</sub>). This will be displayed for each follow-up for both randomized groups.

Table 1: Patient baseline characteristics:

| Characteristics | Neuromuscular exercise and pain neuroscience education group | Pain neuroscience education alone group |
|---|---|---|
| Age (years), mean (SD) | | |
| Sex (men/women, n, %) | | |
| Height (cm), mean (SD) | | |
| Body mass (kg), mean (SD) | | |
| Body mass index (kg/m²), mean (SD) | | |
| Average daily pain intensity<br>over last week (numerical rating<br>scale), mean (SD) | | |
| Index knee (left/right, n, %) | | |
| Dominant leg (left/right, n, %) | | |
| Time since surgery (months), mean (SD) | | |
| Total knee arthroplasty in non-<br>index knee (yes/no, n, %) | | |
| Comorbidities* (n, %) | | |
| The Hospital Anxiety and<br>Depression Scale (0-21), mean<br>(SD) | | |

<sup>\*</sup> The following comorbidities will be recorded: Osteoarthritis in other areas than the index knee, chronic pain from other sites than the index knee, chronic obstructive pulmonary disease, diabetes, and cardiovascular disease.

# **Section 6: Analysis**

### **Outcome definitions**

Item 26: Specification of outcome and timings

Table 2 specifies which outcomes are collected, the timepoints for their assessment and the analysis methods. Further details can be found in the open access protocol (1).

Table 2: Overview of primary, secondary and other outcomes. For more details, please refer to the open access protocol (1)

| | Instrument for assessment | Timing of assessment | Analysis method |
|---|---|---|---|
| Primary outcome – reported in primary publication | | | |

| VOOS man value of | VOOS subsectes asia susuateurs | Danalina 2 6 12 | D |
|---|---|---|---|
| KOOS <sub>4</sub> , mean value of four KOOS subscales | KOOS subscales pain, symptoms, | Baseline, 3-, 6-, 12-, and 24-months | Repeated measures |
| | activities of daily living and knee- | and 24-monus | mixed model |
| scores | related quality of life | | illixed illodel |
| | Each question in KOOS is assigned a | | |
| | score from 0 to 4 and a normalized | | |
| | score (100 indicating no symptoms | | |
| | and 0 indicating extreme symptoms) is calculated for each subscale. The | | |
| | KOOS <sub>4</sub> subscales scores are | | |
| | aggregated and averaged as the | | |
| Sacandamy autoomos | primary outcome | | |
| | reported in primary publication | Dagalina 2 6 12 | Damastad |
| KOOS | All KOOS subscales, i.e., pain, | Baseline, 3-, 6-, 12-, | Repeated |
| | symptoms, activity of daily living, | and 24-months | measures |
| | sport/recreation and knee-related | | mixed model |
| C1.1.1 P 1 | quality of life are individually reported | Danilla 2 6 12 | D 1 |
| Global Perceived | Questionnaire | Baseline, 3-, 6-, 12-, | Repeated |
| Effect | | and 24-months | measures |
| 40 4 6 4 | T' 1 1 1 10 1 | D 1: 2 ( 12 | mixed model |
| 40-meter fast-paced | Time to complete the 40-meter | Baseline, 3-, 6-, 12-, | Repeated |
| walk test | walking test and calculation of | and 24-months | measures |
| ~ | walking speed (meters/second) | - 11 a c 14 | mixed model |
| Stair climb test | Time to complete the stair climb test | Baseline, 3-, 6-, 12-, | Repeated |
| | | and 24-months | measures |
| | | | mixed model |
| 30-second chair stand | Number of chair stands in the 30sec. | Baseline, 3-, 6-, 12-, | Repeated |
| test | chair stand test | and 24-months | measures |
| | | | mixed model |
| Usage of pain | Patient self-report of usage of pain | Baseline, 3-, 6-, 12-, | Poisson |
| medication | medication during last week registered | and 24-months | regression |
| | as yes/no. Registration of the number | | model |
| | of Paracetamols (1 gram) and | | |
| | Ibuprofen and other non-steroidal anti- | | |
| | inflammatory drugs (400 mg.). If any | | |
| | additional pain medication was used, | | |
| | this will be registered as well | | |
| • | ted in primary publication | T | |
| Adverse events | Number of adverse events self- | Continuously during | Poisson |
| | reported by the patients and observed | the intervention | regression |
| | by the physiotherapists supervising the | period | model |
| | interventions | | |
| TT '4 1 A ' 4 1 | | D 1' | <b>N</b> T |
| Hospital Anxiety and | Questionnaire. Reported as a baseline | Baseline | No statistical |
| Depression Scale | characteristic | D 1: 0 6 10 | analysis |
| Other treatments | Patient self-report of other types of | Baseline, 3-, 6-, 12-, | Poisson |
| received | treatment received, defined as | and 24-months | regression |
| | treatments that the patient had initiated | | model |
| | because of the index knee (e.g., | | |
| | acupuncture, manual therapy, surgery, | | |
| | physiotherapy) | | |
| Secondary outcomes – | reported in secondary publications | | |

| PainDETECT | Questionnaire | Baseline, 3-, 6-, 12-, | Repeated |
|---|---|---|---|
| | | and 24-months | measures |
| | | | mixed model |
| Fear-avoidance Beliefs | Questionnaire | Baseline, 3-, 6-, 12-, | Repeated |
| Questionnaire – | | and 24-months | measures |
| Physical Activity | | | mixed model |
| Pain Catastrophizing | Questionnaire | Baseline, 3-, 6-, 12-, | Repeated |
| Scale | | and 24-months | measures |
| | | | mixed model |
| Pain intensity in | Average daily pain intensity over the | Baseline, 3-, 6-, 12-, | Repeated |
| various situations | last week, maximal pain intensity | and 24-months | measures |
| | during rest (day and night), stair | | mixed model |
| | climbing, and walking using a | | |
| | numerical rating scale | | |
| Pain location | Number of painful sites concerning | Baseline, 3-, 6-, 12-, | Repeated |
| | habitual pain areas using a pain | and 24-months | measures |
| | drawing on an anatomical body chart | | mixed model |
| Pressure pain | Measured using a handheld algometer | Baseline, 3-, 6-, 12-, | Repeated |
| thresholds | (Somedic, Hörby Sweden) locally at | and 24-months | measures |
| | the index knee and extrasegmentally at | | mixed model |
| | the forearm | | |
| Conditioned pain | Measured using pressure pain | Baseline, 3-, 6-, 12-, | Repeated |
| modulation | threshold as test stimuli and a spring- | and 24-months | measures |
| | based pressure clamp as conditioning | | mixed model |
| | stimuli | | |
| Pinprick hyperalgesia | Measured locally at the index knee and | Baseline, 3-, 6-, 12-, | Repeated |
| | extrasegmentally at the forearm using | and 24-months | measures |
| | a pinprick nylon filament (Chicago | | mixed model |
| | Medical Supply) | | |
| Temporal summation | Measured locally at the index knee and | Baseline, 3-, 6-, 12-, | Repeated |
| | extrasegmentally at the forearm using | and 24-months | measures |
| | a pinprick nylon filament (Chicago | | mixed model |
| D : 1 : | Medical Supply) | D 1: 2 ( 12 | D . 1 |
| Dynamic mechanic | Measured locally at the index knee and | Baseline, 3-, 6-, 12-, | Repeated |
| allodynia | extrasegmentally at the forearm using | and 24-months | measures |
| D .: | a cotton swab | D 1: 2 ( 12 | mixed model |
| Deep somatic | Measured locally at the index knee and | Baseline, 3-, 6-, 12-, | Repeated |
| hyperalgesia | extrasegmentally at the forearm using | and 24-months | measures |
| Maximal lan aytanaian | a pressure algometer (syringe) | Dogalina 2 6 12 | mixed model |
| Maximal leg extension | Measured in Watt using a leg | Baseline, 3-, 6-, 12-, | Repeated |
| power | extension power rig (Nottingham | and 24-months | measures<br>mixed model |
| | power rig, Nottingham, UK) for index and non-index knee | | mixed model |
| Maximal isometric | Measured in Newton using a handheld | Racalina 2 6 12 | Repeated |
| muscle strength of | dynamometer (Lafayette Manual | Baseline, 3-, 6-, 12-, and 24-months | Repeated measures |
| knee extensors and | Muscle Tester, Loughborough, UK or | and 24-monus | mixed model |
| flexors | MicroFET2, Hoggan Scientific, LLC, | | mixed model |
| HCAUIS | Salt Lake City UT, USA | | |
| | Calculation of isometric | | |
| | hamstring/quadriceps (H/Q) ratio for | | |
| | index and non-index knee using the | | |
| | formula "isometric hamstring strength | | |
| | Tormala isometric namstring strength | l | |

| divided with isometric quadriceps |
|-----------------------------------|
| strength = H/Q ratio" |

KOOS: Knee injury and Osteoarthritis Outcome Score.

## **Analysis methods**

#### Item 27:

Primary, pre-specified secondary and other outcomes presented in table 2 will be reported in the primary 12-month follow-up publication. The same outcomes will be presented for the secondary publication of long-term follow-up when the 24-month data collection is completed (approximately March 2024). Remaining secondary outcomes presented in table 2 will be presented in subsequent, secondary publications.

The primary outcome will be the between-group change in KOOS4 from baseline to 12-month follow-up. Statistical tests will be dependent on data distribution. Validation of normal distribution will be done by reviewing data frequency in histograms and tests for normality (Shapiro-Wilk). For continuous outcomes, we expect data to be normally distributed, and therefore, will be using a repeated measures mixed model with patients as random effect and visit (baseline, 3-, 6-, 12-months) and treatment arm (neuromuscular exercises and pain neuroscience education or pain neuroscience education alone) as fixed effects, and with adjustment for baseline imbalance. Interaction between follow-up and treatment arm was also included in the models. Both crude and adjusted values will be reported.

Secondary outcomes will be analyzed like the primary outcome as well as the long-term (24-month) follow-up analysis. Frequency of adverse events and other types of treatment received (see table 2) will be compared between-groups at the 12-months follow-up using a Poisson regression model with a robust error variance(18). Similarly, between-group comparison of relative risks concerning usage of pain medication will be analyzed using a Poisson regression model, with robust error variance.

A confidence interval including 10 points or more for the primary outcome KOOS<sub>4</sub> will be interpreted as a clinical meaningful difference.

A responder analysis, illustrating the proportion of patients in each randomized group that experienced a minimal clinically important improvement (i.e., minimum improvement of 10 points) for the primary outcome KOOS<sub>4</sub>, will be made to evaluate between-group difference baseline to 12-months follow-up. Results will be analyzed using a Chi-squared test.

A figure including data from all time points (baseline, 3-, 6-, and 12-months) will be presented to visualize the mean value and 95% CI over time in KOOS4 for the patients randomized to either neuromuscular exercise and pain neuroscience education or pain neuroscience education alone. A similar figure will be displayed for the secondary, long-term (24-months) follow-up analysis including all time points (baseline, 3-, 6-, 12-, and 24-months)

The patient's individual trajectory of pain (illustrated by the KOOS pain subscale) and physical performance (illustrated by the 40-meter fast-paced walk test) will be depicted in graphs for both

randomized groups in the subsequent, secondary 12-months follow-up publications and for the secondary long-term (24-month) follow-up publication.

#### Missing data:

Item 28:

Since the linear mixed effects models includes all patients when at least the baseline value or a follow-up value is present, no imputation will be required (19,20). Number of data points available in each group at baseline, 3-, 6-, and 12-months will be displayed in primary and secondary publications. Number of data points available in each group at baseline, 3-, 6-, 12-, and 24-months will be displayed in in the secondary long-term follow-up (24-months) publication.

#### Additional analyses

Item 29:

Exploratory analyses of associations between pre-specified outcomes are planned and will be reported in secondary publications.

Multivariate linear regression models based on the enter method with an adjustment for age, sex, and BMI will be conducted to analyze associations between the primary outcome (KOOS<sub>4</sub>) and pain-related outcomes, bedside quantitative sensory testing outcomes and physical performance outcomes. Two regression models will be conducted. One will include KOOS<sub>4</sub> as the dependent variable and leg extension power and maximal isometric muscle strength for knee flexors and extensor as independent variables and one will include KOOS<sub>4</sub> as the dependent variable and pressure pain thresholds, temporal summation, the fear-avoidance beliefs questionnaire and the pain catastrophizing questionnaire as independent variables.

An exploratory analysis is planned and will be reported in a secondary publication. All patients will be stratified according to their conditioned pain modulation responses, i.e., classified as a conditioned pain modulation responder, a conditioned pain modulation non-responder or no change in conditioned pain modulation. Further details for the stratification are described in the study Larsen et al. Stratification of facilitatory or inhibitory conditioned pain modulation responses in patients with chronic knee pain. Explorative analysis from a multicenter trial (under review at European Journal of Pain). Following stratification, data will be analyzed like the primary analysis (item 27). This analysis will allow us to verify if the treatment effect for the primary and secondary outcomes at 12-months is associated with conditioned pain modulation responses. Results will be presented with a figure including all data points (baseline, 3-, 6-, and 12-months) to visualize the mean and 95% CI over time for the primary outcomes KOOS4 for each randomized group, stratified according to the conditioned pain modulation responses.

Further exploratory analyses can be conducted if deemed relevant.

#### Harms

Item 30: Sufficient detail provided on summarizing harms

Adverse events that may have occurred during the trial period will be identified by the patients (self-reported) and by the physiotherapists supervising the interventions (observations) (see table 3).

Adverse events are characterized as occurring in either the index knee or sites other than the index knee and serious events are defined according to the definitions from the U.S. Food and Drug Administration(21). Adverse events will be descriptively summarized for each randomized group similar to table 3 and be reported in the primary 12-months follow-up publication.

Table 3: Adverse events. The table will include all serious and non-serious adverse events that were registered during the 12-month follow-up period. Serious adverse events associated with the interventions is defined as events that result in death, a life-threating condition, hospitalization, disability or permanent damage, or other serious events, that does not fit the other outcomes (21).

| Adverse events | Neuromuscular exercise and pain neuroscience education group | Pain neuroscience education alone group |
|---|---|---|
| | Number of events | |
| Serious events | | |
| Site other than index knee: | | |
| XXXX | | |
| XXXX | | |
| XXXX | | |
| Index knee: | | |
| XXXX | | |
| XXXX | | |
| XXXX | | |
| All serious events | | |
| Non-serious events* | | |
| Sites other than index knee | | |
| XXXX | | |
| XXXX | | |
| XXXX | | |
| <u>Index knee</u> | | |
| XXXX | | |
| XXXX | | |
| XXXX | | |
| All non-serious | | |

| events |
|--------|

<sup>\*</sup> Non-serious adverse events could be, but not limited to, increased pain in index knee, swelling of index knee, decreased range of motion, distortion of joints, musculoskeletal pain.

#### Statistical software

Item 31: Details of statistical package used for the analysis

The statistical package StataCorp. 2021. Stata Statistical Software: Release 17. College Station, TX: StataCorp LLC was used for data management and analysis. The packages basetable and matrixtools were also used.

#### References

Item 32: Data management

The project is approved by The Danish Data Protection Agency (Aalborg University, 2018-899/10-0166). Data are stored in accordance with the stipulations in The Danish Personal Data Protection Act and other relevant Danish legislation. Data was recorded in hard copy during the outcome assessments and thereafter noted in Excel spreadsheets. Data entry and coding of the non-personal information will be administered by trained staff from Aalborg University. The main data set will not contain any personal information. No personal information will be shared outside the study group. All data, including hard copy data from the individual outcome assessment of the patients, will be stored securely.

The analyses described in this SAP will be the basis of all primary and secondary endpoints. Analyses will be made by the same independent statistician. The principal investigator will code the randomized groups in "group A" and "group B" before submitting the dataset to the statistician. Thereby, analyses will be blinded towards treatment allocation. First, the dataset will be provided for the statistician without information of adherence or adverse events to avoid that blinding is broken. Following finalization and reporting of the intention-to-treat analysis, the statistician will be given information on adherence and adverse events to conduct the per-protocol analysis.

To avoid the risk of misleading interpretation, the blinded results from the intention-to-treat analysis (group A vs. group B) will be presented to all authors. The author group will then decide on two different interpretations of the results, one in which group A refer to neuromuscular exercises and pain neuroscience education, and one in which group A refer to pain neuroscience education alone. The interpretations will be registered in a document titled "NEPNEP trial: Blinded data analyses statement of interpretation". Following written registration and agreeing that no further changes will be made, the randomization code is broken, and the correct interpretation can be chosen(22).

## 7. Reference list

1. Larsen JB, Skou ST, Arendt-Nielsen L, Simonsen O, Madeleine P. Neuromuscular exercise and pain neuroscience education compared with pain neuroscience education alone in patients with chronic

- pain after primary total knee arthroplasty: study protocol for the NEPNEP randomized controlled trial. Trials. 2020 Feb 24;21:218. <a href="https://doi.org/10.1186/s13063-020-4126-5">https://doi.org/10.1186/s13063-020-4126-5</a>
- 2. Peat G, McCarney R, Croft P. Knee pain and osteoarthritis in older adults: a review of community burden and current use of primary health care. Ann Rheum Dis. 2001 Feb;60(2):91–7.
- 3. Dieppe PA, Lohmander LS. Pathogenesis and management of pain in osteoarthritis. Lancet. 2005;365(9463):965–73.
- 4. Hunter DJ, Bierma-Zeinstra S. Osteoarthritis. Lancet. 2019 Apr 27;393(10182):1745–59.
- 5. Price AJ, Alvand A, Troelsen A, Katz JN, Hooper G, Gray A, et al. Knee replacement. Lancet. 2018 Nov 3;392(10158):1672–82.
- 6. Wylde V, Beswick A, Bruce J, Blom A, Howells N, Gooberman-Hill R. Chronic pain after total knee arthroplasty. EFORT Open Rev. 2018 Aug 16;3(8):461–70.
- 7. Rice DA, Kluger MT, McNair PJ, Lewis GN, Somogyi AA, Borotkanics R, et al. Persistent postoperative pain after total knee arthroplasty: a prospective cohort study of potential risk factors. Br J Anaesth. 2018 Oct;121(4):804–12.
- 8. Beswick AD, Wylde V, Gooberman-Hill R, Blom A, Dieppe P. What proportion of patients report long-term pain after total hip or knee replacement for osteoarthritis? A systematic review of prospective studies in unselected patients. BMJ Open. 2012 Feb 22;2(1):e000435.
- 9. Wylde V, Dieppe P, Hewlett S, Learmonth ID. Total knee replacement: is it really an effective procedure for all? Knee. 2007 Dec;14(6):417–23.
- 10. Wright A, Moss P, Sloan K, Beaver RJ, Pedersen JB, Vehof G, et al. Abnormal quantitative sensory testing is associated with persistent pain one year after TKA. Clin Orthop Relat Res. 2015 Jan;473(1):246–54.
- 11. Phillips JR, Hopwood B, Stroud R, Dieppe PA, Toms AD. The characterisation of unexplained pain after knee replacement. Br J Pain. 2017 Nov;11(4):203–9.
- 12. Eitner A, Hofmann GO, Schaible HG. Mechanisms of Osteoarthritic Pain. Studies in Humans and Experimental Models. Front Mol Neurosci. 2017 Nov 3;10:349.
- 13. Roos EM, Lohmander LS. The Knee injury and Osteoarthritis Outcome Score (KOOS): from joint injury to osteoarthritis. Health Qual Life Outcomes. 2003 Nov 3;1:64.
- 14. Skou ST, Roos EM, Laursen MB, Rathleff MS, Arendt-Nielsen L, Simonsen O, et al. A Randomized, Controlled Trial of Total Knee Replacement. N Engl J Med. 2015 Oct 22;373(17):1597–606.
- 15. The European Agency for the Evaluation of Medicinal Products C. Points to consideron multiplicity issues in clinical trials. EMEA. 2002;
- 16. Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361–70.
- 17. Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, et al. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c869.

- 18. Zou G. A modified poisson regression approach to prospective studies with binary data. Am J Epidemiol. 2004 Apr 1;159(7):702–6.
- 19. Ranstam J, Turkiewicz A, Boonen S, van Meirhaeghe J, Bastian L, Wardlaw D. Alternative analyses for handling incomplete follow-up in the intention-to-treat analysis: the randomized controlled trial of balloon kyphoplasty versus non-surgical care for vertebral compression fracture (FREE). BMC Med Res Methodol. 2012 Mar 24;12:35.
- 20. Twisk JW, Rijnhart JJ, Hoekstra T, Schuster NA, ter Wee MM, Heymans MW. Intention-to-treat analysis when only a baseline value is available. Contemp Clin Trials Commun [Internet]. 2020 Dec 1 [cited 2023 Jan 10];20. Available from: https://pubmed.ncbi.nlm.nih.gov/33319119/
- 21. US Food and DA. What is a serious adverse event? [Internet]. Vol. 2018. 2016. Available from: https://www.fda.gov/Safety/MedWatch/HowToReport/ucm053087.htm
- 22. Järvinen TLN, Sihvonen R, Bhandari M, Sprague S, Malmivaara A, Paavola M, et al. Blinded interpretation of study results can feasibly and effectively diminish interpretation bias. J Clin Epidemiol [Internet]. 2014 Jul 1 [cited 2022 Dec 7];67(7):769–72. Available from: http://www.jclinepi.com/article/S0895435613004861/fulltext